CLINICAL TRIAL: NCT07118579
Title: Effects of Remimazolam and Ciprofol Total Intravenous Anesthesia on Perioperative Respiratory Adverse Events in Pediatric Tonsillectomy and Adenoidectomy: A Randomized Controlled Study
Brief Title: Effects of Remimazolam and Ciprofol TIVA on PRAE in Pediatric Tonsillectomy and Adenoidectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RCTIVA
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Tonsillectomy With or Without Adenoidectomy
Keywords: Remimazolam; Ciprofol; TIVA; PRAE
MeSH Terms: interventions — remimazolam; Propofol; (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol group (Active Comparator): Anesthesia induction (2-3 mg/kg) + Anesthesia maintenance (6-10 mg/kg/h)
  Interventions: Drug: Propofol
- Remimazolam group (Experimental): Anesthesia induction (0.3-0.5 mg/kg) + Anesthesia maintenance (1-3 mg/kg/h)
  Interventions: Drug: Remimazolam
- Ciprofol group (Experimental): Anesthesia induction (0.4-0.5 mg/kg) + Anesthesia maintenance (0.8-1.2 mg/kg/h)
  Interventions: Drug: Ciprofol

INTERVENTIONS:
Drug: Remimazolam — remimazolam induction (0.3-0.5 mg/kg) + maintenance (1-3 mg/kg/h)
  Other Names: Remi
  Arms: Remimazolam group
Drug: Propofol — Anesthesia induction (2-3 mg/kg) + Anesthesia maintenance (6-10 mg/kg/h)
  Other Names: PRO
  Arms: Propofol group
Drug: Ciprofol — Anesthesia induction (0.4-0.5 mg/kg) + Anesthesia maintenance (0.8-1.2 mg/kg/h)
  Other Names: CIP
  Arms: Ciprofol group

SUMMARY:
To observe the effects of remimazolam versus ciprofol TIVA on PRAE in pediatric tonsillectomy and adenoidectomy.

DETAILED DESCRIPTION:
To observe the effects of remimazolam versus ciprofol TIVA on PRAE in pediatric tonsillectomy and adenoidectomy, aiming to enhance surgical safety and improve postoperative outcomes in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2-12 years
* ASA physical status I-II
* Body mass index (BMI): 14-28 kg/m²
* Scheduled for elective tonsillectomy with or without adenoidectomy
* Signed informed consent by legal guardian(s) and assent by children (≥8 years old)

Exclusion Criteria:

* History of severe pulmonary diseases (e.g., asthma, bronchiectasis, severe OSA)
* Previous episodes of significant PRAEs
* Documented drug allergies (e.g., to remimazolam, propofol, or ciprofol)
* Comorbidities including: Uncorrected congenital heart disease, neuromuscular disorders, Developmental delay, Abnormal hepatic/renal function
* Preoperative moderate-to-severe respiratory infections requiring surgery postponement
* Recent participation in other clinical trials

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of perioperative respiratory adverse events | 5days
  The perioperative respiratory adverse events including: laryngospasm, bronchospasm, severe cough, oxygen desaturation, airway obstruction.

SECONDARY OUTCOMES:
Anesthesia duration | 1 day
  From anesthesia induction to discontinuation of anesthetics
Emergence time | 1 day
  From anesthetic discontinuation to eye opening on command
Extubation time | 1 day
  From anesthetic discontinuation to endotracheal tube removal
PACU stay duration | 1 day
  From PACU admission to meeting discharge criteria
The modified Aldrete score | 1 day
  Upon admission to the PACU, the child was assessed using the modified Aldrete score, which ranges from 0 to 10. A higher score indicates a better recovery status.
doses of drugs | 24 hours
  Total sedative/analgesic consumption

CONTACTS AND LOCATIONS:
Overall Officials: Mujun Chang, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No